CLINICAL TRIAL: NCT00378547
Title: Effect of Paracetamol Versus Paracetamol Combined With Pregabalin Versus Paracetamol Combined With Pregabalin and Dexamethasone on Pain and Opioid Requirements in Patients Scheduled for Tonsillectomy
Brief Title: Effect of Paracetamol, Pregabalin and Dexamethasone on Pain and Opioid Requirements in Patients Having a Tonsillectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: ENT surgery stopped at the recruiting hospital
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Ole Mathiesen, Section of Acute Pain Management and Palliative Care
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM4-05
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Pain, Postoperative
Keywords: Tonsillectomy; pregabalin; dexamethasone; multimodal postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Pregabalin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paracetamol (Placebo Comparator): Oral paracetamol 1 g + placebo + placebo
  Interventions: Drug: paracetamol + placebo + placebo
- Paracetamol + Pregabalin (Experimental): Oral paracetamol 1g + oral pregabalin 300 mg + placebo
  Interventions: Drug: paracetamol + pregabalin + placebo
- Paracetamol + pregabalin + dexamethasone (Experimental): Oral paracetamol 1g + oral pregabalin 300 mg + IV dexamethasone 8 mg
  Interventions: Drug: paracetamol + pregabalin + dexamethasone

INTERVENTIONS:
Drug: paracetamol + placebo + placebo — Comparing the analgesic effect of combinations of paracetamol + placebo + placebo
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: paracetamol + pregabalin + placebo — Comparing the analgesic effect of combinations of paracetamol + pregabalin 300 mg + placebo
  Other Names: Acetaminophen; Pregabalin
  Arms: Paracetamol + Pregabalin
Drug: paracetamol + pregabalin + dexamethasone — Comparing the analgesic effect of combinations of paracetamol + pregabalin 300 mg + dexamethasone 8 mg
  Other Names: Acetaminophen; Pregabalin; Dexamethasone
  Arms: Paracetamol + pregabalin + dexamethasone

SUMMARY:
Patients scheduled for a tonsillectomy need postoperative pain treatment. Some of the most widely used postoperative analgetics (NSAIDs) sometimes cause rebleeding in the postoperative period, and another often used analgetic, morphine, causes nausea and vomiting. The researchers therefore will investigate new combinations of postoperative analgesics in hopes of improving pain and the need for opioids during the postoperative period.

DETAILED DESCRIPTION:
We will investigate the effect of paracetamol versus paracetamol combined with pregabalin versus paracetamol combined with pregabalin and dexamethasone on pain and morphine requirements in the first 24 hours postoperatively. Outcomes include amount of morphine and ketobemidone used, and pain measured on a VAS scale. Side-effects, e.g., PONV, dizziness and sedation are also measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for benign tonsillectomy
* Between the ages of 18 and 50 years old
* ASA 1-2 and a surgical technique without the need for local anaesthetics or electrical scissors

Exclusion Criteria:

* Malignancy
* Patients who are unable to cooperate
* Does not speak Danish
* Has allergy for drugs used in the trial
* Has abused drugs and/or medicine
* Epilepsy
* Diabetes treated with medicine
* Treatment with systemic steroids 4 weeks prior to the operation
* Daily use of antacids
* Daily use of analgesics
* Use of antidepressives
* Known kidney disease
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain score (VAS) 2, 4, and 24 hours postoperatively. | 0-24 hours
Both at rest and when swallowing 50 ml of water. | 0-24 hours

SECONDARY OUTCOMES:
Total amount of morphine and ketobemidone used 0-24 hours postoperatively. | 0-24 hours
Nausea and vomiting 2, 4, and 24 hours postoperatively. | 0-24 hours
Dizziness and sedation 2, 4, and 24 hours postoperatively. | 0-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, Study Chair — Department of Anaesthesiology, Copenhagen University Hospital in Glostrup, 2600 Glostrup, Denmark
Locations (1):
- Department of Day Case Surgery at Glostrup University Hospital, Glostrup Municipality, Denmark